CLINICAL TRIAL: NCT05038605
Title: Topical Versus Oral Metronidazole for Pain Relief After Surgery for Benign Anorectal Conditions; a Prospective Randomized Study
Brief Title: Topical vs Oral Metronidazole After Benign Anorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Associate professor of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mansoura2021
Record Dates: First submitted 2021-08-29; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Hemorrhoids; Anal Fissure; Anal Fistula
MeSH Terms: conditions — Hemorrhoids; Fissure in Ano; Rectal Fistula | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical metronidazole (Active Comparator): Topical application of metronidazole cream on the anal verge after surgery
  Interventions: Drug: Topical metronidazole
- Oral metronidazole (Active Comparator): oral metronidazole 500 mg tablets after surgery
  Interventions: Drug: oral metronidazole
- Control (No Intervention): No metronidazole was received

INTERVENTIONS:
Drug: Topical metronidazole — Topical application of metronidazole cream on the anal verge every 8 hours after surgery
  Arms: Topical metronidazole
Drug: oral metronidazole — Patients received oral metronidazole 500 mg tablets every 8 hours after surgery
  Arms: Oral metronidazole

SUMMARY:
While some investigators found oral metronidazole to be effective in reducing pain after hemorrhoidectomy, other researchers did not find a significant analgesic effect of systemic metronidazole. On the other hand, topical application of metronidazole had more consistent favorable results as Ala et al documented a remarkable analgesic effect of topical metronidazole 10% after excisional hemorrhoidectomy which was in line with Nicholson and Armestrong who also concluded similar results.

No previous study compared the analgesic effect of topical and oral metronidazole after anorectal surgery. Therefore, the present trial was conducted to compare the impact of oral versus systemic metronidazole on pain and recovery after surgery for benign anorectal conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex aged below 70 years
* Underwent surgery for hemorrhoids, anal fissure, or simple anal fistula.

Exclusion Criteria:

* Grade I-II hemorrhoids.
* acute anal fissure.
* complex anal fistula
* perianal abscess
* perianal Crohn's disease
* malignancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score | at one day after surgery
  Pain was assessed using visual analogue scale form 0 to 10, higher score indicates worse pain
Postoperative pain score | at two days after surgery
  Pain was assessed using visual analogue scale form 0 to 10, higher score indicates worse pain
Postoperative pain score | at seven days after surgery
  Pain was assessed using visual analogue scale form 0 to 10, higher score indicates worse pain

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No